CLINICAL TRIAL: NCT00771628
Title: Comparison of Flex-It Stylet to Malleable Stylet for GlideScope Intubation: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other); Unity Health Toronto (Other)
Responsible Party: Timothy Turkstra, University of Western Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-08-111; 13949
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Intubation
Keywords: Intubation, Flex-It, stylet, GlideScope

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flex-It Stylet (Experimental): Patients will be intubated using the GlideScope with an ETT fitted with a Flex-It stylet.
  Interventions: Device: Flex-It Stylet
- 2 Malleable (Active Comparator)
  Interventions: Device: Standard malleable stylet

INTERVENTIONS:
Device: Flex-It Stylet — Patients will be intubated using the GlideScope with an ETT fitted with a Flex-It stylet.
  Arms: Flex-It Stylet
Device: Standard malleable stylet — Patients will be intubated using the GlideScope with an ETT fitted with a standard malleable stylet.
  Arms: 2 Malleable

SUMMARY:
Patients presenting for elective surgery requiring tracheal intubation will be randomized to one of two different ETT stylets. The primary outcome is time to intubation.

The null hypothesis is that there will be no difference.

The GlideScope video laryngoscope (Verathon) is a widely used intubating device that uses a high-resolution camera embedded into a plastic laryngoscope blade. An LED provides illumination. The GlideScope often provides a good laryngoscopic view, but passing the endotracheal tube (ETT) through the vocal cords is sometimes difficult. Because of the 60 degree anterior curvature of the GlideScope's blade, ETT's must have stylets inserted so that the ETT distal tip can be positioned anteriorly. Various authors have recommended different angles of the ETT to optimally place it into the trachea, including matching the GlideScope's 60 degree angle, or configuring the ETT with a 90 degree bend. Previous studies demonstrated that 90 degree sharp bend was both faster and subjectively easier in a heterogeneous group of intubators. With the introduction of the Flex-It stylet by Parker Medical, the question arises as to the the best configuration of stylet for the ETT. Therefore, this prospective, randomized, single-blinded trial is proposed.

DETAILED DESCRIPTION:
Written informed consent will be obtained by one of the study investigators, and a copy will be given to each participant. Written informed consent will also be obtained from the operator of the GlideScope. Envelopes with computer-generated randomized group assignments will be present at each site. The envelopes will be consecutively numbered (i.e. "U1", "U2" for University Hospital, "S1", "S2" for St Joseph's Health Care, etc.). After consent, randomization will occur by selecting the next consecutive envelope. The envelope will contain the data collection form as well as a piece of paper that has the following information:

* at the top will be the randomization group (A, B) and a text description of the endotracheal tube angle and stylet (i.e. "90 degrees - malleable stylet")
* in the body of the piece of paper will be a template that shows the exact shape into which the tube must be bent, including where the distal and proximal ends are, the angle of curvature that must be followed, and the location along the length of the tube at which to create this angle. The angle and location will be the same for both males and females.

There are three distinct anesthesia providers involved in the conduct of this study, as follows:

1. "operator" - person performing the intubation
2. "timer" - person timing the outcome (one of the co-investigators)
3. "shaper" - person who ensures that the angle and stylet of the tube matches the group to which the patient was allocated

Because the person intubating must be blind up until the time at which the tube is to be used, the unopened envelope will be taken to a third anesthesia provider, who will prepare the ETT with stylet in an area that is not visible to the person performing the intubation or to the person timing the intubation. The person performing the intubation will specify what size of tube to be prepared. This will most commonly be 7.5 mm internal diameter (ID) for a female and 8.0 ID for males, but the operator is free to use whatever size they feel is appropriate. The tube size selection will take place before unblinding so the group allocation cannot affect the decision of tube size.

The tubes will all be cut at the 27 cm marking. "Group A" ETT's will be shaped with the aid of a standard malleable stylet (Rusch 14 Fr) that has been lubricated with single-use water-soluble lubricant. "Group B" ETT's will be instrumented with the Flex-It Stylet, with identical lubricant. The prepared tube will then be concealed under a standard green OR towel and brought to the operating room (OR). This tube will be placed close to the patient's head so that it is readily accessible.

Data Collection

In the OR, the GlideScope will be turned on at least 60 seconds before use so that the lens can warm-up to prevent fogging. The patient will be cared for in the usual fashion with respect to monitoring and induction of general anesthesia. To ensure adequate pre-oxygenation, the patient's end-tidal oxygen must be ≥ 70%. Muscle relaxation will be used, and the agent used is at the discretion of the operator. After induction of anesthesia, bag-mask ventilation will be used in the usual fashion until the operator decides to proceed to laryngoscopy with the GlideScope. The operator will remain blinded to the group allocation until after the laryngoscopic view has been obtained with the GlideScope, where upon he will be handed the endotracheal tube.

The timer (who cannot see the tube under the green towel) will watch the operator until the GlideScope is inserted into the patient's mouth, start the timer, and then turn 180º to face the anesthetic monitor. The timer will not be able to see the ETT, stylet, or curvature because he will be facing the monitor screen.

Timing will continue until end-tidal CO2 of at least 30 mmHg is seen on the anesthesia monitor, at which point the data collection form will be filled out, and the study protocol will be finished. (The time to intubation will be recorded to the nearest tenth of a second.) If the operator fails to intubate within 3 attempts or 150 seconds, the intubation will be noted as a failure, and the ultimately successful means of securing the airway will be recorded.

The definition of an "attempt" for the purposes of this clinical trial are as follows:

1. anytime the GlideScope blade is removed from the patients mouth and then re-inserted
2. anytime the endotracheal tube is re-shaped (regardless of whether or not the GlideScope is actually removed from the patient's mouth
3. if substantial adjustments are made to the patient's position (such as head position, neck flexion, or neck extension). Small movements that would occur in the normal process of intubation would not count as "substantial".

If oxygen desaturation (as recorded by pulse oximetry) below 95% occurs, then the patient will be ventilated in the usual fashion to ensure oxygenation, and re-attempting intubation using the GlideScope may proceed, but the timing will continue, and the same limits to successful intubation (within 3 attempts or total of 150s) will apply. Between attempts, the tube may be re-shaped by the operator if the operator feels that another curvature would be preferred.

ELIGIBILITY:
Inclusion Criteria:

1. * Any adult patient scheduled for elective surgery.
2. ETT is indicated for the procedure in the opinion of the attending anesthesiologist.
3. Any operator who has performed ≥ 10 GlideScope intubations.

Exclusion Criteria:

1. Any patient in whom the use of the GlideScope is contraindicated in the opinion of the attending anesthesiologist.
2. * Patient with known cervical spine abnormalities.
3. * Any patients with known or probable difficult airways (this rare occurrence is unlikely to be evenly distributed between the groups and could skew the data).
4. Any patient requiring rapid sequence induction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Time to Intubation | Prospective 10-150 seconds

SECONDARY OUTCOMES:
Ease of Intubation Visual Analog Scale | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Turkstra, MD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

REFERENCES:
- [Derived] Turkstra TP, Jones PM, Ower KM, Gros ML. The Flex-It stylet is less effective than a malleable stylet for orotracheal intubation using the GlideScope. Anesth Analg. 2009 Dec;109(6):1856-9. doi: 10.1213/ANE.0b013e3181bc116a. PMID 19923515